CLINICAL TRIAL: NCT06958094
Title: Effectiveness of Gamified Mobile Health Apps for Airway Clearance Therapy in Children and Adolescents With Cystic Fibrosis: A 24-Week Randomized Controlled Trial.
Brief Title: Effectiveness of Gamified Mobile Health Apps for Airway Clearance Therapy in Children and Adolescents With Cystic Fibrosis
Acronym: EGmACT-CF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Córdoba (Other)
Responsible Party: Principal Investigator, Alvaro Alba Rueda, Prof, Universidad de Córdoba
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAFQFISIO2025
Record Dates: First submitted 2025-04-27; First posted 2025-05-06 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Cystic Fibrosis (CF)
Keywords: MHealth; Gamification; Mobile App; Adherence; Engagement; Motivation; Children; Adolescent; Randomized Controlled Trial
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental Group (Experimental): At least twelve participants will engage in airway clearance therapy using gamified mobile health (mHealth) applications. These apps are designed to promote the control of sound intensity during open-glottis expiratory maneuvers, utilizing the smartphone's integrated microphone to detect vocal output. The sound generated during breathing reflects active respiratory effort and effective glottic control, supporting secretion mobilization and enhancing airway clearance efficacy.
  Interventions: Other: Gamified mobile health applications
- Control Group (Active Comparator): At least twelve participants will undergo treatment with conventional airway clearance techniques. These techniques are designed to promote effective secretion mobilization and improve lung function. Participants will be guided through a series of controlled breathing exercises aimed at optimizing airflow and enhancing secretion clearance. These methods involve active participation to perform specific maneuvers that facilitate the removal of mucus from the airways, improving overall respiratory function.
  Interventions: Other: Conventional Airway Clearance Therapy
- Mixed Intervention Group (Active Comparator): At least twelve participants will undergo a combined intervention, consisting of 10 minutes of gamified mHealth app use followed by 10 minutes of conventional airway clearance techniques, or the sequence may be reversed. This dual approach will enable participants to benefit from both interactive digital engagement and established respiratory therapies, optimizing mucus clearance and enhancing overall pulmonary function.
  Interventions: Other: Combination Treatment

INTERVENTIONS:
Other: Gamified mobile health applications — * Voice Volume Catcher: A game where players control a character's movement by modulating their voice volume. Louder or softer sounds move a basket to collect different types of fruits, encouraging continuous vocal engagement and fine control of breath intensity.
  * Scream Go Hero: A voice-controlled platform game where players produce short or long vocalizations to make the hero character jump or move across obstacles. The game demands breath control and supports prolonged exhalations for larger jumps with an open glottis, which is beneficial for airway clearance.
  * Chicken Scream: A voice-activated game where players guide a chicken character by varying their vocal intensity to make it walk, jump, and avoid enemies. Participants must dynamically adjust their breath pressure and vocal intensity while maintaining open-glottis breathing, promoting agility in respiratory control.
  Other Names: Gamified mHealth Apps
  Arms: Experimental Group
Other: Conventional Airway Clearance Therapy — * Autogenic Drainage: A technique where participants perform a series of controlled breathing cycles-deep inhalations followed by forceful exhalations-to mobilize mucus from the lower airways to the upper airways. The technique encourages breath control and helps clear secretions without the need for coughing, promoting efficient airway clearance.
  * Active Cycle of Breathing Techniques (ACBT): In this technique, participants alternate between relaxed breathing, deep breaths, and huffing to mobilize and expel mucus from the lungs. It focuses on breathing control to loosen and expel secretions effectively while maintaining a steady airflow throughout the process.
  * Positive Expiratory Pressure (PEP) Therapy: This technique involves exhaling against a resistance through a device, which helps to open the airways and prevent their collapse. The resistance promotes prolonged exhalations, facilitating the movement of mucus from the small airways to the larger airways for easier clearance.
  Arms: Control Group
Other: Combination Treatment — - Gamified mHealth Apps (10 minutes):
  Voice Volume Catcher
  Scream Go Hero
  Chicken Scream
  - Conventional Airway Clearance Techniques (10 minutes):
  Autogenic Drainage
  Active Cycle of Breathing Techniques (ACBT)
  Positive Expiratory Pressure (PEP) Therapy
  Arms: Mixed Intervention Group

SUMMARY:
The aim of this randomized controlled trial is to evaluate the effectiveness of gamified mobile health (mHealth) applications for airway clearance therapy in children and adolescents with cystic fibrosis. Primary outcomes include Forced Vital Capacity (FVC), Forced Expiratory Volume in the first second (FEV₁), adherence to therapy, health-related quality of life (HRQoL), and satisfaction with the intervention. The intervention will consist of 20-minute sessions, performed twice daily over a 24-week period. At least a total of 36 participants aged 8 to 18 years with cystic fibrosis will be randomly assigned to three equally sized groups: the experimental group (gamified mHealth apps: Voice Volume Catcher, Scream Go Hero, and Chicken Scream), the control group (conventional airway clearance techniques: Autogenic Drainage, Active Cycle of Breathing Techniques, and Positive Expiratory Pressure therapy), and the mixed group (10 minutes of gamified mHealth apps combined with 10 minutes of conventional techniques). This study seeks to provide evidence on the feasibility and clinical benefits of integrating gamification into airway clearance therapy to improve respiratory outcomes and patient engagement in pediatric cystic fibrosis care.

ELIGIBILITY:
* Inclusion Criteria:

  * Population with cystic fibrosis (CF), aged 8-20 years.
  * Individuals using or not using CFTR modulators (e.g., Kaftrio, Kalydeco, etc.), regardless of their specific mutation.
* Exclusion Criteria:

  * Forced Vital Capacity (FVC) and/or Forced Expiratory Volume in the first second (FEV1) < 40%.
  * Oxygen therapy or continuous mechanical ventilation.
  * Moderate hemoptysis or recent pneumothorax (within the past 3 months).
  * Presence of an active, uncontrolled respiratory infection exacerbation that required hospitalization within the 30 days prior to the intervention.
  * Other conditions such as neuromuscular disorders or cognitive difficulties (Mini-Mental State Examination score < 19 points).

Ages: 8 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Forced Vital Capacity (FVC) | This outcome will be measured at three points: baseline, 12 weeks, and 24 weeks.
  Total volume of air that can be forcibly exhaled after a full inhalation. It is a key parameter measured during spirometry testing to assess lung function.
Forced Expiratory Volume in the first second (FEV₁) | This outcome will be measured at three points: baseline, 12 weeks, and 24 weeks.
  The volume of air exhaled during the first second of a forced exhalation after a full inhalation. It is a key parameter measured during spirometry testing to assess airflow and diagnose respiratory conditions.
Adherence to therapy | This outcome will be measured at three points: baseline, 12 weeks, and 24 weeks.
  The extent to which participants follow the prescribed therapeutic regimen. Adherence will be assessed over time using the gamified mHealth app (experimental group), a stopwatch application (control group), or a combination of both (mixed intervention group), all monitored through the StayFree app.
Health-related quality of life (HRQoL) | This outcome will be measured at three points: baseline, 12 weeks, and 24 weeks.
  This measure will evaluate the impact of cystic fibrosis on participants' daily lives, including physical, emotional, and social well-being. The age-adapted Cystic Fibrosis Questionnaire-Revised (CFQ-R) will be used. The CFQ-R scores range from 0 to 100, with higher scores indicating better health-related quality of life. Cut-off points may vary depending on the study's context, but scores below 50 are often interpreted as indicating significant impairment in quality of life.
Satisfaction with the intervention | This outcome will be measured at three points: baseline, 12 weeks, and 24 weeks.
  The outcome will be assessed using the Treatment Satisfaction Questionnaire for Medication (TSQM), adapted for a physical therapy intervention. This tool will measure participants' contentment with the therapy and their overall treatment experience. The TSQM scores range from 0 to 100 for each domain (effectiveness, side effects, convenience, and global satisfaction), with higher scores indicating greater satisfaction. There are no universally established cut-off points, but higher scores typically reflect more positive treatment experiences.

CONTACTS AND LOCATIONS:
Locations (1):
- Asociación Andaluza de Fibrosis Quística, Seville, Seville, Spain